CLINICAL TRIAL: NCT06396910
Title: Immune Maping of Tuberculosis and Sarcoidosis Granuloma
Brief Title: TB and Sarcoidosis Granuloma
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Martin Rottenberg, Professor, Karolinska Institutet
Other Study IDs: 2021-03760
Record Dates: First submitted 2024-04-30; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Tuberculosis; Sarcoidosis
MeSH Terms: conditions — Tuberculosis; Sarcoidosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Paraffin blocks of lung tissues obtained for diagnostic purposes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Spatial transcriptomics — Localize immune transcripts in the pulmonary lessions of sarcoidosis and tuberculosis patients. This is done in biopsies from pathological libraries.

SUMMARY:
Tuberculosis (TB) and sarcoidosis are both granulomatous diseases. Here we compared the immunological micro-environments of granulomas from TB and sarcoidosis patients using in situ sequencing (ISS) transcriptomic analysis and multiplexed immunolabelling of tissue sections.

DETAILED DESCRIPTION:
Tuberculosis (TB) and sarcoidosis are diseases that are characterized by the formation of inflammatory structures called granulomas. TB is caused by infection with the bacteria Mycobacterium tuberculosis while sarcoidosis is a an inflammatory disease of unknown ethiology. We hypothesize that the localization of immune molecules in granulomas determines the the course of TB and sarcoidosis using in situ sequencing, a spatial transcriptomic technology and immunolabelling in biopsies from patients. In the project, we aim to answer the following questions: 1. How does the immune landscape differ in different TB granulomas (with/without necrosis, different histology)? 2. How does the immune landscape differ in acute (Lofgren's syndrome) and chronic (non-Lofgren's syndrome) sarcoidosis samples? 3. How does the immune landscape differ in histologically similar granulomas from TB and sarcoidosis patients? We will use in situ sequencing that can identify the exact location of 65 specific immune markers in the lung at the same time, thereby correlating defined immune landscapes with the histology, bacterial content and disease type.

ELIGIBILITY:
Inclusion Criteria:

Specimen were taken from patients with a confirmed diagnosis of TB based on granulomatous inflammation based on histopathological confirmation together with additional parameters such as, clinical symptoms, radiological and laboratory parameters (microscopy detection of acid-fast bacilli in sputum, M. tuberculosis culture, chest radiography, and MTB/RIF GeneXpert analysis) were included.

Sarcoidosis and TB biopsies were selected by a clinical patholologist that evaluated the ocurrence of the granulomatous lessions

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We utilized retrospective historical samples of patients either with TB or sarcoidosis from the Aga Khan University Hospital Clinical Laboratories, Karachi, Pakistan (TB: n=10), the BioMaterialBank North, Research Center Borstel, Germany (sarcoidosis, n=7; TB=1) and the Karolinska University Hospital (Sarcoidosis, n=4). The FFPE samples used were originally obtained for diagnostic purposes.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Spatial transcriptome of lung lesions of sarcoidosis and tuberculosis patients | 14 days
  We will detect individual mRNA molecules in patietn lessions with cellular definition and retaining the positional information

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carow B, Muliadi V, Skalen K, Yokota C, Kathamuthu GR, Setiabudiawan TP, Lange C, Scheu K, Gaede KI, Goldmann T, Pandita A, Masood KI, Pervez S, Grunewald J, Hasan Z, Levin M, Rottenberg ME. Immune mapping of human tuberculosis and sarcoidosis lung granulomas. Front Immunol. 2024 Feb 7;14:1332733. doi: 10.3389/fimmu.2023.1332733. eCollection 2023. PMID 38385142